CLINICAL TRIAL: NCT06061692
Title: Tongxinluo Capsule in the Treatment of Cerebral Small Vessel Disease-A Randomized, Double-blind, Placebo-controlled, Multicenter Clinical Study (TOPS-CSVD)
Brief Title: Tongxinluo Capsule in the Treatment of Cerebral Small Vessel Disease-A Randomized, Double-blind, Placebo-controlled, Multicenter Clinical Study（TOPS-CSVD）
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Qiang Dong, Chief physician, Huashan Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TOPS-CSVD
Record Dates: First submitted 2023-09-25; First posted 2023-09-29 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Cerebral Small Vessel Diseases
Keywords: Cerebral Small Vessel Diseases, cognitive impairment
MeSH Terms: conditions — Cerebral Small Vessel Diseases; Cognitive Dysfunction | interventions — tongxinluo

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test group (Experimental): Tongxinluo Capsule, 4 capsules/time, tid, p.o
  Interventions: Drug: Tongxinluo Capsule
- Control group (Placebo Comparator): Tongxinluo Capsule placebo, 4 capsules/time, tid, p.o
  Interventions: Drug: Tongxinluo Capsule

INTERVENTIONS:
Drug: Tongxinluo Capsule — 4 capsules/time, tid, p.o Duration of Treatment: 1 year (12 months)

SUMMARY:
Cerebral small vessel disease is a series of clinical, imaging and pathological syndromes caused by various etiologies affecting the arteries, capillaries, venules in the brain. The common causes of cerebral small vessel disease include arteriolosclerosis, cerebral amyloid angiopathy, hereditary cerebral small vessel disease, inflammation-and immune-mediated small vessel disease, venous collagen disease and other small vessel diseases. Of these, age-and hypertension-related cerebral small vessel disease and amyloidosis cerebral small vessel disease are the most common types. The pathophysiological mechanism and clinical manifestations of cerebral small vessel disease are complex. One-fifth of ischemic strokes and the vast majority of nontraumatic parenchymal hemorrhages are due to cerebral small vessel disease. In addition to stroke, patients with cerebral small vessel disease are more often characterized by chronic progressive neurological impairment, which is an important cause of cognitive decline and functional disability in the elderly, and has become one of the important public health problems affecting the quality of life of the elderly.

Focusing on cognitive impairment-related diseases, a large number of clinical studies have shown that Tongxinluo capsule has a dual neurovascular protective effect, which can increase the Mini-Mental State Examination (MMSE) score and activities of daily living (ADL) score of patients with lacunar cerebral infarction combined with vascular cognitive impairment, reduce fibrinogen (FIB) concentration, improve whole blood viscosity, improve blood viscosity and FIB level, improve activities of daily living and accelerate intellectual recovery in patients with VD; It can also reduce the levels of ET-1 and homocysteine in AD patients, reduce the whole blood viscosity and thus improve the microcirculation in the elderly, increase cerebral blood flow, increase the scores of MMSE and ADL, improve the intelligence of patients, improve memory disorders and language disorders. Meta-analysis of 3458 patients in 40 published clinical literatures of Tongxinluo capsule both domestically and internationally confirmed that Tongxinluo capsule had the effect of promoting the recovery of neurological function, and was safe without adverse reactions.

This project is a randomized, double-blind, placebo-controlled multicenter clinical study to investigate the clinical efficacy and safety of Tongxinluo capsule in the treatment of cerebral small vessel disease. A total of 1052 subjects who met the subject screening criteria are planned to be enrolled, with 526 patients in the test group and 526 patients in the placebo group.

The study is conducted using a central randomization method. For the patients who met the inclusion criteria after examination, they are logged into the Interactive Web Response System by their site, entered the relevant information, and randomized and assigned drugs automatically by the central server according to the ratio of 1:1. Once enrolled, all patients receive the study drug (Tongxinluo or placebo) at 4 capsules/tid for up to 12 months. The study is planned to be conducted at approximately 50 centers across the country using central randomized competing enrollment.

ELIGIBILITY:
Inclusion Criteria:

1. Age 50-80 years (both inclusive);
2. Complaints of cognitive impairment involving memory and/or other cognitive domains for at least 3 months;
3. Neither normal nor demented cognitive level according to DSM-V criteria, MMSE scale score ≥20 (elementary school) or ≥24 (junior high school and above); CDR scale score ≥0.5 in at least one domain and overall CDR score ≤1;
4. MRI has: ① moderate to severe white matter lesions (deep Fazekas score > 1 or paraventricular Fazekas score > 2); Mild white matter hyperintensity (deep Fazekas score = 1 or paraventricular Fazekas score = 2) combined with more than 1 lacunar infarction or more than 3 microbleeds foci. ② Absence of old cortical or watershed infarction, cerebral hemorrhage, hydrocephalus, and other cerebral white matter lesions of definite etiology (e.g., multiple sclerosis, metabolic, toxic, etc.);
5. Voluntary participation in the study and willing to sign the Informed Consent Form.

Exclusion Criteria:

1. Previously diagnosed with dementia;
2. Acute stroke event within 6 months;
3. Previously diagnosed hereditary or inflammatory small vessel disease;
4. Presence of congenital mental retardation and severe neurological and psychiatric diseases;
5. Illiterate or severe visual or hearing impairment that may prevent patients from cooperating with neuropsychological assessment;
6. Relevant depression (Hamilton Depression Scale score ≥ 17 points), or other unrelated serious mental illness (schizophrenia, bipolar disorder or delirium);
7. Combined with severe cardiac, pulmonary and renal insufficiency (creatinine > 2.0 mg/dL or 177 μmol/L), severe hepatic impairment (transaminase more than 3 times of normal value);
8. Alcohol abuse, drug abuse or use of drugs affecting cognitive assessment, such as sedatives, hypnotics, nootropic drugs, cholinergic drugs;
9. Definitely diagnosed malignant tumor, vital organ failure;
10. Previous allergy or intolerance to Tongxinluo ingredients;
11. The subject has no stable and reliable caregiver, or the caregiver is unable to help the subject participate in the whole process of the study;
12. Patients who have participated in other interventional clinical studies within the last 3 months, or are participating in other interventional clinical studies.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1052 (Estimated)
Dates: Start 2023-10 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Changes in Vascular Dementia Cognitive Assessment Scale (VADAS-cog) at 1 year. | 1 year
  Changes in Vascular Dementia Cognitive Assessment Scale (VADAS-cog)

SECONDARY OUTCOMES:
Incidence rate of combined endpoint at 1 year: including new stroke (ischemic [TOAST classification] or hemorrhagic)/transient ischemic attack, myocardial infarction, new dementia and death; | 1 year
  Incidence rate of combined endpoint at 1 year: including new stroke (ischemic [TOAST classification] or hemorrhagic)/transient ischemic attack, myocardial infarction, new dementia and death;
The incidence rate of each individual event of the combined endpoint at 1 year; | 1 year
  The incidence rate of each individual event of the combined endpoint
Changes in Clinician Interview-Based Impression of Change Scale (CIBIC-Plus) at 1 year; | 1 year
  Changes in Clinician Interview-Based Impression of Change Scale (CIBIC-Plus)
Change from baseline in Mini-Mental State Examination (MMSE) at 1 year; | 1 year
  Change from baseline in Mini-Mental State Examination (MMSE)
Change from baseline in Symbol Digit Modalities Test (SDMT) at 1 year; | 1 year
  Change from baseline in Symbol Digit Modalities Test (SDMT)
Change from baseline in Clinical Dementia Rating Scale (CDR) at 1 year; | 1 year
  Change from baseline in Clinical Dementia Rating Scale (CDR)
Change from baseline in Neuropsychiatric Inventory Questionnaire (NPI-Q) at 1 year; | 1 year
  Change from baseline in Neuropsychiatric Inventory Questionnaire (NPI-Q)
Change from baseline in Activity of Daily Living Scale (ADL) at 1 year; | 1 year
  Change from baseline in Activity of Daily Living Scale (ADL)
Change from baseline in motor score (TUG, 3-meter walking time) at 1 year; | 1 year
  Change from baseline in motor score (TUG, 3-meter walking time)

OTHER OUTCOMES:
Volume changes in brain regions at 1 year; | 1 year
  Volume changes in brain regions
Volume changes in cerebral white matter at 1 year; | 1 year
  Volume changes in cerebral white matter
Changes in number of cerebral microbleeds at 1 year; | 1 year
  Changes in number of cerebral microbleeds
Changes of cerebral blood flow at 1 year. | 1 year
  Changes of cerebral blood flow.

IPD SHARING:
Plan to Share IPD: No
The IPD will not share for confidentiality reasons

REFERENCES:
- [Derived] Wang Y, Xie X, Xu J, Lei P, Wang K, Zhang J, Yu J, Cui M, Dong Q. Tongxinluo capsule in the treatment of cerebral small vessel disease: protocol of a randomised, double-blind, placebo-controlled, multicentre clinical study (TOPS-CSVD). Stroke Vasc Neurol. 2025 Sep 10:svn-2024-003929. doi: 10.1136/svn-2024-003929. Online ahead of print. PMID 40935402